CLINICAL TRIAL: NCT06861569
Title: Effect of Positive End-expiratory Pressure on the Gastric Volume in Patients Undergoing General Anesthesia with Supraglottic Airway Device: a Prospective Randomized Controlled Non-inferiority Trial
Brief Title: Effect of Positive End-expiratory Pressure on the Gastric Volume
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, BON WOOK KOO, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: SNUBH-LMASONOPEEP
Record Dates: First submitted 2025-02-15; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-04

CONDITIONS: Gastric Volume; Breast Cancer Female; Anesthesia Complication
Keywords: Supraglottic Airway Device; Postive End Expiratory Pressure; Gastric Sonography
MeSH Terms: interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ZEEP (No Intervention): Patients undergoing general anesthesia using supraglottic airway device without PEEP.
- PEEP (Experimental): Patients undergoing general anesthesia using supraglottic airway device with PEEP of 5cmH2O.
  Interventions: Procedure: Positive end expiratory pressure

INTERVENTIONS:
Procedure: Positive end expiratory pressure — Positive end-expiratory pressure (PEEP) is a value that can be set up in patients receiving invasive or non-invasive mechanical ventilation. 5cmH2O PEEP will be applied to the PEEP group participants.
  Arms: PEEP

SUMMARY:
The main purpose of this study is to quantitatively evaluate the effect of applying PEEP during the use of SGA on gastric volume, aiming to provide objective evidence regarding the potential side effects, such as gastric volume increase. It is expected that this will contribute to improving the quality of patient management through the safe clinical use of SGA and PEEP.

DETAILED DESCRIPTION:
General anesthesia has positive effects in relieving pain and unpleasant memories during surgery by blocking the patient's voluntary movements and reflexes to stimuli. However, it can lead to side effects such as severe impairment or absence of spontaneous breathing, necessitating artificial respiration. Among the conventional airway management methods for artificial respiration, the supraglottic airway device (SGA) has the advantage of reducing hemodynamic changes, intracranial pressure, and intraocular pressure caused by airway stimulation, as it does not pass through the airway, and it reduces airway-related complications. However, a disadvantage is its inability to adequately seal the airway, making it difficult to use in cases where there is a high risk of aspiration or when high airway pressures are required.

Positive End Expiratory Pressure (PEEP) has the advantage of preventing atelectasis, improving oxygen exchange capacity, and preventing pulmonary complications by maintaining lung expansion. However, applying PEEP increases airway pressure, and if the SGA does not adequately seal the airway, there is a possibility of air entering the stomach. If air enters the stomach and increases gastric volume, the risk of postoperative vomiting and aspiration pneumonia increases due to increased gastric pressure. Also, increased intra-abdominal pressure and diaphragmatic elevation can lead to respiratory distress due to decreased lung volume during postoperative recovery.

While there are studies suggesting that PEEP can be safely used with SGA, there is a need for verification as there are no studies objectively measuring changes in gastric volume using methods such as ultrasound when using PEEP with SGA. The main purpose of this study is to quantitatively evaluate the effect of applying PEEP during the use of SGA on gastric volume, aiming to provide objective evidence regarding the potential side effects, such as gastric volume increase. It is expected that this will contribute to improving the quality of patient management through the safe clinical use of SGA and PEEP.

Before entering the operating room, patients will be placed in a sitting and right lateral decubitus (RLD) position to measure the cross sectional area(CSA) of the stomach antrum using ultrasound. One investigator will scan the sagittal plane in the upper abdominal region using a low-frequency ultrasound probe (2-5 MHz) and measure the major diameter (D1) and transverse diameter (D2) of the observed antrum. CSA can be calculated from the measured values as in formula (a) below. The investigator will scan three times for each posture, and calculate the average.

CSA = D1 x D2 x 1/4 ------- (a) Using CSA, gastric volume (GV) is estimated using formula (b) below. GV (ml) = 27.0 + 14.6 × CSA - 1.28×age ------- (b) Midazolam premedication is not administered before surgery. When patients enter the operating room, standard monitoring devices (electrocardiogram, pulse oximetry, non-invasive blood pressure monitor, BIS or SedLine) are attached for vital sign monitoring, and target-controlled infusion of propofol is initiated at a target concentration of 4.0 µg/ml, and remifentanil at a target concentration of 3.0 ng/ml.

After confirming loss of consciousness and loss of spontaneous respiration, SGA is inserted, and the position of the SGA is evaluated and recorded using the fiberoptic scoring system.

During surgery, maintenance of anesthesia is managed with target-controlled infusion of propofol to keep BIS (Bispectral Index) between 40-60 or PSI (Patient State Index) between 25-49. For adequate analgesia during surgery, remifentanil is continuously infused using target-controlled infusion.

At 5 minutes (T0), 30 minutes (T1), and 60 minutes (T2) after SGA insertion, the following values related to mechanical ventilation are measured: FiO2 (Fraction of Inspired Oxygen), PIP (Peak Inspiratory Pressure), RR (Respiratory Rate), lung compliance, SpO2 (Oxygen Saturation), EtCO2 (End-tidal Carbon Dioxide), TV (Tidal Volume), OLP (Oropharyngeal Leak Pressure), leak volume, and leak fraction.

Immediately after surgery, CSAright-lat and GV are measured as described in above. After confirming that respiration and consciousness levels have returned to clinically normal conditions post-surgery, the patient is discharged to the recovery room, and assessments are made for nausea or vomiting, respiratory depression, sore throat, and blood staining.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 19 and above.
* Patients scheduled for general anesthesia for elective surgery.
* American society of anesthesiologists physical status classification 1 or 2

Exclusion Criteria:

* Individuals who have not provided prior consent for participation in the study
* Patients showing cognitive impairment to the extent that voluntary consent is difficult
* Obesity with a BMI of 30 kg/m² or higher
* Patients with anatomical abnormalities in the airway structure making supraglottic airway device application difficult
* Patients with respiratory diseases making PEEP application difficult (e.g., chronic obstructive pulmonary disease, asthma)
* Patients suspected of delayed gastric emptying (e.g., not adhering to fasting guidelines, medication use affecting gastric motility [anticholinergics, narcotic analgesics], neurological disorders [Parkinson's disease, multiple sclerosis], diabetes, hypothyroidism)
* Patients with a history of gastrointestinal surgery
* Pregnant women
* Patients undergoing concurrent surgeries or collaborative procedures
* Patients transferred from the intensive care unit

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Gastric volume difference before and after surgery | Baseline and end of surgery 0 minute
  Before and after the surgery, the patient is positioned in a sitting position and then in the right lateral decubitus (RLD) position. Ultrasound is used to measure the cross-sectional area (CSA) of the gastric antrum and then it is substituted into the following equation to estimate gastric volume.
  GV (ml) = 27.0 + 14.6 × CSAright-lat - 1.28×age The scanning is performed three times for each position to obtain the average value.

SECONDARY OUTCOMES:
Fraction of Inspired Oxygen | 5 minutes, 30 minutes, 60 minutes after SGA insertion
  The measured values during mechanical ventilation are averaged.
Peak Inspiratory pressure | 5 minutes, 30 minutes, 60 minutes after SGA insertion
  The measured values during mechanical ventilation are averaged.
Respiratory rate | 5 minutes, 30 minutes, 60 minutes after SGA insertion
  The measured values during mechanical ventilation are averaged.
Lung compliance | 5 minutes, 30 minutes, 60 minutes after SGA insertion
  The measured values during mechanical ventilation are averaged.
Oxygen Saturation | 5 minutes, 30 minutes, 60 minutes after SGA insertion
  The measured values during mechanical ventilation are averaged.
End-tidal carbon dioxide | 5 minutes, 30 minutes, 60 minutes after SGA insertion
  The measured values during mechanical ventilation are averaged.
Tidal volume | intraoperative period
  The measured values during mechanical ventilation are averaged.
Oropharyngeal leak pressure | 5 minutes, 30 minutes, 60 minutes after SGA insertion
  The measured values during mechanical ventilation are averaged.
Leak volume and leak fraction | 5 minutes, 30 minutes, 60 minutes after SGA insertion
  The measured values during mechanical ventilation are averaged. Leak volume is defined as the difference between inspired and expired tidal volume. Leak fraction is defined as the ratio of leak volume/inspired tidal volume.
Presence of blood staining on SGA | Immediately after the end of anesthesia
  When the SGA is removed after the surgery, check whether there is blood staining on the SGA.
The duration of stay in the recovery room after surgery | upto 1 hour after entering the recovery room
  The time from admission to the recovery room to discharge
Presence of postoperative nausea and vomiting | upto 1 hour after entering the recovery room
  Postoperative nausea and vomiting which occur during the time from the end of surgery until discharge from the recovery room.
Presence of respiratory depression | upto 1 hour after entering the recovery room
  Respiratory depression which occurs during the time from the end of surgery until discharge from the recovery room.
Presence of sore throat | upto 1 hour after entering the recovery room
  Sore throat which occurs during the time from the end of surgery until discharge from the recovery room.

CONTACTS AND LOCATIONS:
Overall Officials: Bon Wook Koo, Study Chair — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol